CLINICAL TRIAL: NCT06743841
Title: Study of the Efficacy of a New Nutritional Supplement, Compared with Placebo, in Promoting Active and Healthy Aging from the Age of 65
Brief Title: Study of a Nutritional Supplement for Healthy Aging
Acronym: ACTIPRO SENIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTIPRO SENIOR (2021.116)
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Nutrition, Healthy; Quality of Life
Keywords: Healthy aging; Nutritional status; Nutritional supplement; Quality of life
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: A randomized, parallel, double-blind, 8-week nutritional intervention trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional Supplement (Experimental): 1 sachet of nutritional supplement (30g) in the morning and 1 sachet (30g) in the afternoon during 8 weeks. A total of 60g daily.
  Interventions: Dietary Supplement: Nutritional supplement
- Control (Placebo Comparator): 1 sachet of placebo supplement (30g) in the morning and 1 sachet (30g) in the afternoon during 8 weeks. A total of 60g daily.
  Interventions: Dietary Supplement: Control supplement

INTERVENTIONS:
Dietary Supplement: Nutritional supplement — 60g of a nutritional supplement powder, divided into 2 daily intakes, one in the morning and one in the afternoon
  Arms: Nutritional Supplement
Dietary Supplement: Control supplement — 60g of a placebo supplement powder, divided into 2 daily intakes, one in the morning and one in the afternoon
  Arms: Control

SUMMARY:
The main aim of this clinical trial is to learn if a nutritional supplement improves health status from a nutritional point of view in an active and healthy elderly population. It will also study about the improvement of anthropometric variables, vitality, quality of life and mood, as well as biochemical and metabolic changes produced after the intervention.

The main questions it aims to answer are:

* Does a nutritional supplement improve the general nutritional status?
* What health parameters improve most clearly after taking the supplement? Researchers will compare a nutritional supplement to a placebo (a look-alike substance that contains no interest nutrients) to see if the nutritional supplement works to improve health status from a nutritional point of view.

Participants will:

* Take a nutritional supplement or a placebo every day for 8 weeks.
* Visit the clinic once every 4 weeks for checkups and tests
* Keep a diary of their symptoms and the degree of adherence to taking the nutritional supplement.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 65 and 80 years of age, inclusive.
* Body mass index (BMI) less than 35 kg/m2.
* Subjects must have a cultural level, general physical and psychological conditions that allow the understanding, monitoring and development of the study.
* Agree to voluntarily participate in the study and provide their informed consent in writing, complying with the procedures and requirements of the study.

Exclusion Criteria:

* People allergic to soy or lactose, as the supplement contains traces.
* Severe diseases or relevant functional or structural abnormalities of the digestive system: inflammatory bowel disease.
* Surgical interventions of the digestive system with permanent sequelae such as resections (gastroduodenostomy…)
* Presenting any type of serious or chronic or systemic disease such as: infections that cause impairment of the general condition, cardiovascular diseases, cardiac arrhythmias, stroke, neoplasia, severe kidney disease, liver disease…
* Recent fracture in the last 3 months (strength training).
* Subjects who present some type of cognitive and/or psychological impediment, Alzheimer's, depressive pathology, etc.
* Pharmacological treatment that affects the study variables recently prescribed, without a stable dose prescribed.
* People with diabetes of any type.
* Intake of any type of nutritional supplement that includes vitamin D, folic acid, vitamin B6, vitamin B12, calcium, iron, zinc or proteins, in the last 3 months.
* Being on any type of special diet and/or high alcohol consumption (more than 14 units in women and 20 units in men per week).
* Subjects in whom poor collaboration is expected or who, in the opinion of the researcher, have difficulties in following the procedures of the study.
* Lack of commitment (in the opinion of the researcher) to the intervention, suspicion of non-compliance, or real difficulties in following the development of the study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Nutritional score. | Days 0 and 56
  A nutritional score was created ad hoc to estimate the effects of a nutritional supplement . The parameters included in the score were: muscle mass, lymphocyte level, protein status, vitamin D, folic acid, vitamin B12, calcium, iron, zinc, and homocysteine levels

SECONDARY OUTCOMES:
Dietary intake | Days 0 and 56
  Analysis of dietary intake (types of food and energy and nutritional value of the diet), using a food frequency questionnaire
Height | Days 0 and 56
  Height will be measured by stadiometer and reported in m.
Weight | Days 0 and 56
  Weight will be measured by bioimpedance and reported in kg.
Waist circumference | Days 0 and 56
  Waist circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Hip circumference | Days 0 and 56
  Hip circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Total adipose tissue | Days 0 and 56
  Total adipose tissue will be analyzed by dual-energy x-ray absorptiometry scan and electrical bioimpedance
Visceral adipose tissue | Days 0 and 56
  Visceral adipose tissue will be analyzed by dual-energy x-ray absorptiometry scan and electrical bioimpedance
Lean mass | Days 0 and 56
  Lean mass will be analyzed by dual-energy x-ray absorptiometry scan and electrical bioimpedance
Upper limb strength | Days 0 and 56
  Upper limb strength will be measured in the bench press exercise
Lower limb strength | Days 0 and 56
  Lower limb strength will be measured using the sit-and-stand test in 30 seconds
Maximum hand grip | Days 0 and 56
  Maximum hand grip will be measured using a manual dynamometer
Blood fasting glucose | Days 0 and 56
  Blood will be extracted at fasting state and glucose levels will be determined by autoanalyzer Pentra-C200.
Blood fasting insulin | Days 0 and 56
  Blood will be extracted at fasting state and insulin levels will be determined by ELISA.
Total cholesterol | Days 0 and 56
  Blood will be extracted at fasting state and Total cholesterol levels of participants will be analysed by autoanalyzer Pentra-C200.
HDL-cholesterol | Days 0 and 56
  Blood will be extracted at fasting state and HDL cholesterol levels of participants will be analysed by autoanalyzer Pentra-C200.
LDL-cholesterol | Days 0 and 56
  LDL cholesterol levels of participants will be calculated by Friedewald equation.
Triglycerides | Days 0 and 56
  Blood will be extracted at fasting state and triglyceride levels of participants will be analysed by autoanalyzer Pentra-C200.
C-Reactive Protein | Days 0 and 56
  C-Reactive Protein will be measured in an automated ELISA processing system
Interleukin 6 | Days 0 and 56
  Interleukin 6 will be measured in an automated ELISA processing system
Tumor necrosis factor -α | Days 0 and 56
  Tumor necrosis factor -α will be measured in an automated ELISA processing system
Blood pressure | Days 0 and 56
  Systolic and Diastolic blood pressure in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Depression level | Days 0 and 56
  Depression level will be measured by the validated Spanish translation of the Beck Depression Inventory (BDI)
Anxiety level | Days 0 and 56
  Anxiety level will be measured by by the validated Spanish translation of the State-Trait Anxiety Inventory (STAI)
Short Form-36 questionnaire | Days 0 and 56
  Quality of life is measure by the Short Form -36, a questionnaire with eight scales physical functioning, physical role limitation, pain, general health, vitality, social functioning, emotional role limitations and general health perception

CONTACTS AND LOCATIONS:
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain